CLINICAL TRIAL: NCT05733806
Title: Prospective, Multicenter, Observational Study on Rare Gynecological Cancers
Brief Title: Study on Gynecological Rare Cancers
Acronym: MITO9B
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MITO 9B
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Gynecologic Cancer
Keywords: rare cancers; gynecologic malignancies
MeSH Terms: interventions — Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic rare tumors: The study will include patients with rare gynecologic malignancies
  Interventions: Other: chemotherapy, surgery

INTERVENTIONS:
Other: chemotherapy, surgery — this is an observational prospective study, therefore no intervention is planned. Patients perform medical and surgical treatment as per standard of case.

SUMMARY:
This is a prospective, observational, multicenter study on gynecological rare tumors.

DETAILED DESCRIPTION:
This is a prospective registry aimed to better understand prognosis, clinical and pathological features, management of this rare cancer conditions for improving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* rare gynecological malignancies
* written informed consent
* patient fit for follow-up

Exclusion criteria

-written informed consent not provided

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — patient with gynecologic cancers
Study Population: Patients with rare gynecological malignancies
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gynecologic rare malignancies | 5 years
  To describe the prevalence of gynecologic rare tumors

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, MD, Principal Investigator — IRCCS Fondazione G Pascale, Naples
Locations (2):
- Italy (2):
  - Ginecologia e Ostetricia, IRCCS Ospedale San Raffaele, Milan
  - IRCCS Fondazione G Pascale, Naples

IPD SHARING:
Plan to Share IPD: No